CLINICAL TRIAL: NCT03881813
Title: Effectiveness of Two Types of Fixed Lingual Retainers in Preventing Mandibular Incisor Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Nasreen Iqbal Nagani, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DUHS/DR-0/2017/327
Record Dates: First submitted 2019-03-17; First posted 2019-03-20 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Relapse
Keywords: fixed retainers; alignment
MeSH Terms: conditions — Recurrence | interventions — Orthodontic Retainers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fiber reinforced composite retainers (Experimental): Fiber reinforced composite retainers were inserted in group 1 and were evaluated after every 3 months for a follow up period of 3 months.
  Interventions: Device: Orthodontic retainers
- Multistranded stainless steel retainers (Experimental): Multistranded stainless steel retainers were inserted in group 2 and were evaluated after every 3 months for a follow up period of 3 months.
  Interventions: Device: Orthodontic retainers

INTERVENTIONS:
Device: Orthodontic retainers — Orthodontic retainers were bonded on the lower teeth of the subjects after fixed orthodontic treatment and were evaluated for their effectiveness for the followup of one year.

SUMMARY:
The study evaluates effectiveness of two types of fixed retainers in post orthodontic patients. Half of the subjects are randomly allocated Group 1 retainer (FRC) and other half is given Group 2 retainer (MSW) and followed for a period of one year.

DETAILED DESCRIPTION:
54 subjects were recruited and divided into two groups by random allocation. Consents were obtained . Group 1 received fiber reinforced composite retainer and group 2 received multistranded stainless steel wire retainer. The patients were recalled at every three months interval for a period of 12 months. They were evaluated for number of fractures, failure pattern based on adhesive remnant index and relapse tendency by measuring little's irregularity index.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed fixed appliance orthodontic treatment.
* Subjects who have signed the consent forms.
* Subjects who have accepted the terms and conditions of visiting after every three months for one year.
* Non extraction cases in the mandibular arch with no IPR.
* Patients without caries/ restoration/ fracture on the lower anterior teeth.
* Patients with healthy periodontium with no periodontal disease at that time.

Exclusion Criteria:

* Presence of syndrome or systemic disease.
* Patients taking medications/ drugs.
* Patients with poor oral hygiene.
* Patients with congenitally absent/ missing anterior teeth in the mandibular arch.
* Patients with habit of clenching/ bruxism.
* Patients with history of betel nut chewing.
* Presence of occlusal interferences.

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2017-11-12 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Relapse tendency | 12 months
  It was measured using Little's irregularity index

SECONDARY OUTCOMES:
Bond failure | 12 months
  Number of bond failure was assessed at each visit.
Failure Pattern | 12 months
  Type of failure pattern was assessed based on Adhesive remnant index.

CONTACTS AND LOCATIONS:
Overall Officials: Nasreen Nagani, BDS, Principal Investigator — DUHS
Locations (1):
- Dow University Of Health Sciences, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nagani NI, Ahmed I, Tanveer F, Khursheed HM, Farooqui WA. "Clinical comparison of bond failure rate between two types of mandibular canine-canine bonded orthodontic retainers- a randomized clinical trial". BMC Oral Health. 2020 Jun 29;20(1):180. doi: 10.1186/s12903-020-01167-7. PMID 32600325